CLINICAL TRIAL: NCT03380234
Title: Reducing Exposure to Tobacco Smoke Among Primary School Students - a Cluster Randomised Controlled Trial
Brief Title: A Cluster-RCT of SHS Among Primary School Students
Acronym: SHS-cRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: coshshs
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Secondhand Smoke; Thirdhand Smoke; Smoking
Keywords: Smoking; Secondhand smoke; Thirdhand smoke; Children; Cluster randomised controlled trial
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 8 worksheets and around 15 online quizzes and 30 WhatsApp messages.
  Interventions: Other: Worksheets; Other: Whatsapp messages; Other: Online quizzes
- Control (Other): Control students will receive the following minimal intervention to reduce their intention to smoke and SHS - a leaflet on smoking and SHS published by the Department of Health.
  Interventions: Other: Leaflet

INTERVENTIONS:
Other: Worksheets — Worksheets will be distributed to students for them and their parents to complete together. During the first 3 months, the teachers will distribute 1 worksheet every two weeks to the intervention grades, and 1 worksheet in the 4th and 5th months as boosters. The worksheets will deliver information about tobacco smoke, SHS and THS, inviting students and their family members to complete other interesting tasks together.
  Arms: Intervention
Other: Whatsapp messages — A mobile phone number of this study is also provided on the worksheets, through which participants can receive WhatsApp/WeChat/instant messages (1-2 times every week) designed to encourage behavioural change [15]. They can then forward selected messages to other members of their household, especially smokers.
  Arms: Intervention
Other: Online quizzes — At the end of each worksheet, a QR code is inserted. By scanning this code, students or parents will be invited to answer 2-3 simple quizzes which allow us to assess students' knowledge obtained from the intervention materials and their avoidance of environmental tobacco smoke.
  Arms: Intervention
Other: Leaflet — A leaflet on smoking and SHS published by the Department of Health will be mailed to the control grades.
  Arms: Control

SUMMARY:
This is a school- and family-based prospective trial among Primary/Grade 2-4 (P2-4) students in randomly selected 12 schools in Hong Kong. This study will assess the intervention effects on children's exposure to environmental tobacco smoke (including SHS and THS at home, SHS at home from neighbours and SHS outside home), children's SHS-related knowledge and attitude, intention to smoke, respiratory symptoms, parents' smoking cessation, and family happiness.

DETAILED DESCRIPTION:
Around 12 primary schools in Hong Kong will be randomly selected and recruited and the 3 grades (P2-4) in each of the recruited schools will be randomly allocated to intervention or control arms. After the consenting process and baseline survey, we will conduct a 3-month intervention and then 2-month boosters which include 8 worksheets, around 15 online question quizzes and 30 WhatsApp messages. After 3-month and 6-month follow-up periods, we will assess the differences of children's exposure to environmental tobacco smoke (including SHS and THS at home, SHS at home from neighbours and SHS outside home), children's SHS-related knowledge and attitude, intention to smoke, respiratory symptoms, parents' smoking cessation, and family happiness. According to the results of baseline survey, we will also invite all the students exposed to SHS at home to provide their hair samples before intervention and at the 6th month in order to obtain objective results (hair nicotine measurements).

Aims of this study: (1) To reduce children's exposure to environmental tobacco smoke. (2) To reduce objectively measured exposure to tobacco smoke (hair nicotine) among children who are exposed to SHS at home at baseline. (6-month, laboratory test). (3) To promote SHS-related knowledge and attitudes, and avoidance of SHS among children. (4) To reduce children's intention to smoke. (5) To reduce children's respiratory symptoms. (6) To promote smoking cessation (past 7 days) of parents. (child report) (7) To promote children's perception of family happiness.

ELIGIBILITY:
We will invite all P2-4 students from 12 schools randomly selected from the 100 schools (which watched the performance by Hong Kong Council on Smoking and Health) to participate in this cluster RCT, as they are able to understand simple questionnaires and other self-help intervention materials, yet remain very receptive to intervention activities from our experience.

Inclusion criteria for hair nicotine test:

1) exposed to secondhand smoke at home from smokers inside home in any of the past 7 days; 2) living with at least 1 smoker; 3) Never smoking or using e-cigarettes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3432 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
To reduce children's exposure to environmental tobacco smoke. | 3 and 6-month
  In the 3th and 6th month, students will conduct a survey to assess their exposure to environmental tobacco smoke.

SECONDARY OUTCOMES:
To reduce the hair nicotine levels of students who are exposed to SHS at home at baseline. | 6-month
  At the 6th months, parents will be invited to post their children's hair for laboratory test and identify the change of the nicotine levels (objective measurement) before and after intervention.
To promote SHS-related knowledge and attitudes, and avoidance of SHS among children. | 3 and 6-month
  In the 3th and 6th month, students will conduct a survey to assess their SHS-related knowledge and attitudes, and avoidance of SHS.
To reduce children's intention to smoke. | 3 and 6-month
  In the 3th and 6th month, students will conduct a survey to assess children's intention to smoke.
To reduce children's respiratory symptoms. | 3 and 6-month
  In the 3th and 6th month, students will conduct a survey to assess children's respiratory symptoms.
To promote smoking cessation (past 7 days) of parents. (child report) | 6-month and 12-month3 and 6-month
  In the 3th and 6th month, students will conduct a survey to report their parents' smoking cessation.
To promote children's perception of family happiness. | 3 and 6-month
  In the 3th and 6th month, students will conduct a survey to report their perception of family happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — School of Public Health, the University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No